CLINICAL TRIAL: NCT04096651
Title: Pathophysiology of Gait and Posture in Progressive Supranuclear Palsy
Acronym: Gait-PSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Collaborators: University Hospital Center of Martinique (Other); Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RBM-PAP-2015/19
Record Dates: First submitted 2019-09-06; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Progressive Supranuclear Palsy
Keywords: progressive supranuclear palsy PSP; atypical parkinsonism; gait disorders; neurophysiology; imaging
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PSP Classic (Other): 15 patients with a "classical" form of PSP are recruited to realize all the tests of the multimodal approach.
  Interventions: Other: gait recordings; Other: brain magnetic resonance imaging; Other: oculomotor movement recordings
- Caribbean PSP (Other): 15 patients with a "Caribbean PSP" are recruited to realize all the tests of the multimodal approach.
  Interventions: Other: gait recordings; Other: brain magnetic resonance imaging; Other: oculomotor movement recordings
- Healthy controls (Other): 15 persons with no PSP are recruited to realize all the tests of the multimodal approach.
  Interventions: Other: gait recordings; Other: brain magnetic resonance imaging; Other: oculomotor movement recordings

INTERVENTIONS:
Other: gait recordings — gait recordings
Other: brain magnetic resonance imaging — brain magnetic resonance imaging
Other: oculomotor movement recordings — oculomotor movement recordings

SUMMARY:
The main hypothesis is that the gait and postural deficits in the Caribbean form of PSP may be associated with a dysfunction of the cerebral cortex, as they result from sub-cortical involvement in classical forms. The investigators will characterize the gait and posture with a force platform to collect biomechanical gait parameters, coupled with the kinematic and electromyographic (EMG) study. Then the investigators realize a multimodal imaging study [structural magnetic resonance imaging (MRI) and diffusion tensor imaging (DTI)] that allow us to determine if a correlation can be found between the clinical characteristics of postural control and walking on one hand, and morphological changes and structural MRI changes in cortico-subcortical pathways on the other hand. The study of performance on neuropsychological tests, registration of ocular movements and the analysis of functional cortical activity will complete our multimodal approach. A better understanding of these disorders is expected to propose new drug treatment and rehabilitative strategies.

DETAILED DESCRIPTION:
Progressive supranuclear palsy (PSP) is a rare neurodegenerative disease (6/100 000 inhabitants) characterized by the association of Parkinson's syndrome, a paralysis of the verticality of the gaze and an alteration early balance and walking with the onset of falls during the first year of evolution of the disease. From a neuropathological point of view, it is characterized by a tauopathy with neurodegeneration within the basal ganglia, cerebellum, and midbrain (which includes the mesencephalic locomotor region-MLR).

In the Caribs this pathology is abnormally frequent (incidence over 3 times higher than expected), and represents 1/3 of the total Parkinsonian syndromes. In these patients, cortical pathology predominates leading to different cognitive deficit relative to patients with the classical form of PSP. Conversely, in PSP patients, imaging data suggest a preferential midbrain-thalamocortical pathway dysfunction. Pathophysiological mechanisms causing gait disturbances and postural control presented by these patients remains however not fully elucidated . In patients with Caribbean PSP, of which the clinical features are specific, gait disorders and falls appear later in the course of the disease (2.5 years on average) suggesting perhaps a different physiopathological mechanism. Consequently weak knowledge of the mechanisms involved, none specific treatment is currently available and the taking in therapeutic charge of these disorders rests essentially on a re-educative approach that remains poorly codified.

In this study, gait and balance disorders will be recorded using a force platform, coupled with kinematic study and EMG in patients with classical form of PSP and Caribbean one, and in controls. The functional and anatomy of brain will be examined using a multimodal brain imaging approach (with DTI. Performance in neuropsychological tests and oculomotor movements will also be measured. A comparative and correlation analyses will be performed to assess the link between gait, balance, oculomotor and cognitive performances and brain anatomy, and the differences between subjects groups. Caribbean PSP patients are recruited from Neurology and Physical Medicine and Rehabilitation of University Hospital of Pointe-à-Pitre and Fort de France, Classical PSP patients are be recruited from the Centre d'Investigation Clinique (CIC) of the Pitié-Salpêtrière hospital, and healthy volunteers from both centers.

ELIGIBILITY:
Inclusion Criteria:

* Patient :
* Patients who met the clinical criteria for PSP and Gd-PSP
* Walking and standing alone without assistance
* Patient or responsible third party who received information about the study and who signed the informed consent
* French
* Patients over 40 years
* Clinically detectable eye movement anomaly

Witnesses :

* To be affiliated or beneficiary of social security scheme
* French person
* Major subjects, matched for age (± 3 years) and sex, showing no neurological or psychiatric disease or severe progressive disease
* No Indication against MRI

Exclusion Criteria:

Patient :

* Patient not affiliated with the social security system
* Cognitive impairment: MMSE ≤ 20; FAB ≤ 12
* psychiatric disorders likely to interfere with exploration; severe postural disorders
* MRI not feasible Witnesses
* Not affiliated or benificiary of social security scheme
* Not a french person
* Somebody showing neurological or psychiatric disease or severe progressive disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
gait velocity | at inclusion
  gait recordings

SECONDARY OUTCOMES:
brain anatomy | at inclusion
  magnetic resonance imaging
oculomotor movements recordings | at inclusion
  oculomotor movements recordings

CONTACTS AND LOCATIONS:
Overall Officials: Annie LANNUZEL, PU-PH, Study Director — University Hospital of Guadeloupe; Régine EDRAGAS, PH, Principal Investigator — University Hospital of Martinique; Marie-Laure WELTER, PU-PH, Principal Investigator — Groupe Hospitalier Pitie-Salpetriere

IPD SHARING:
Plan to Share IPD: No